CLINICAL TRIAL: NCT05322629
Title: Stepped Care to Optimize PrEP Effectiveness in Pregnant and Postpartum Women (SCOPE-PP) in South Africa
Brief Title: Stepped Care to Optimize PrEP Effectiveness in Pregnant and Postpartum Women
Acronym: SCOPE-PP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Cape Town (Other)
Responsible Party: Principal Investigator, Dvora Joseph Davey, PhD, MPH, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-21-1770; 3R01HD106862-04S1 (NIH)
Record Dates: First submitted 2022-03-24; First posted 2022-04-12 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-05

CONDITIONS: Hiv
Keywords: pregnant; postpartum; prevention of mother to child transmission; PrEP; pre-exposure prophylaxis; HIV prevention; breastfeeding
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Breast Feeding

STUDY DESIGN:
Intervention Model Description: In a randomized control trial of 750 women, the study team will evaluate: (1) PrEP continuation (missing <1 PrEP collections) and (2) PrEP adherence per drug levels of TFV-DP at 6m follow up.
  Pregnant women who are on PrEP or initiate PrEP at baseline visit will be recruited and screened for eligibility during their routine antenatal services at gestational >25 weeks using a set script for screening and a brief description of the study. Study staff will obtain written informed consent immediately following screening.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (enhanced PrEP HIV biofeedback) (Experimental): Women in the intervention arm (n=375) will receive enhanced PrEP bio-feedback adherence counseling:
  * Real-time novel immunoassay using urine that measures tenofovir and enhanced bio-feedback counseling. The novel urine assay shows tenofovir concentrations if PrEP is taken in the past 48 hours thereby enabling counselors to provide feedback on adherence levels, immediately.
  * Enhanced counseling on recent adherence levels
  * Rapid PrEP collection
  In second randomization at 6m, women on PrEP with poor adherence or continuation, will be offered differentiated PrEP delivery in the community or in the clinic. The study will follow these participants for 15m to assess longer term PrEP continuation and adherence.
  Interventions: Behavioral: PrEP adherence biofeedback
- Standard of care (Active Comparator): Women in the standard of care arm (n=375) will receive facility-based PrEP and monthly HIV testing in pregnancy and quarterly in postpartum. PrEP prescriptions and HIV testing will be provided according to the national PrEP guidelines. The women will be followed through 6m postpartum for the first randomization and through 15m with the standard of care for the second randomization.
  Interventions: Behavioral: Standard of care counseling

INTERVENTIONS:
Behavioral: PrEP adherence biofeedback — Services for women in the intervention arm includes bio-feedback adherence counseling based on urine lateral flow assays of tenofovir to measure adherence with rapid PrEP delivery .
  Arms: Intervention (enhanced PrEP HIV biofeedback)
Behavioral: Standard of care counseling — Adherence counseling based on self report and following national guidelines
  Arms: Standard of care

SUMMARY:
To reach HIV-uninfected pregnant and breastfeeding women in South Africa, who are at very high risk of HIV, researchers will test a new and innovative package of interventions: 1) pre-exposure prophylaxis (PrEP), which is a daily antiretroviral pill that is both safe and effective for preventing HIV in pregnant and breastfeeding mothers and 2)) enhanced adherence counseling combined with differentiated deliver of community PrEP delivery for women who have difficulties with regular PrEP use.

Our study will be among the first ever to evaluate the efficacy and cost-effectiveness of a PrEP intervention among pregnant and postpartum women and will play a key role in informing maternal PrEP interventions to eliminate HIV acquisition and transmission to partners and their infants.

DETAILED DESCRIPTION:
HIV incidence doubles during pregnancy and postpartum period compared with non-pregnant women, underscoring the urgent need for prevention interventions tailored to high-risk pregnant and breastfeeding women. Incident maternal HIV infections lead to an estimated one-third of all infant HIV infections. South Africa expects over 90,000 infant HIV cases in the next decade; one-third of those can be prevented by eliminating maternal HIV acquisition. Pre-exposure prophylaxis (PrEP) in pregnancy and breastfeeding is safe and effective at preventing HIV. However, PrEP use remains low in pregnancy, and drop precipitously in the postpartum period.

Researchers will test a novel strategy to optimize PrEP in pregnant and postpartum women in South Africa. Our randomized control trial (RCT) is designed to address key barriers to maternal PrEP use and evaluate cost-effectiveness to inform national policy. This trial builds on our earlier work demonstrating the acceptability, feasibility, safety and potential efficacy of a package of interventions including PrEP, enhanced adherence counseling combined with community, differentiated delivery of PrEP for women who want to take PrEP but have difficulties with adherence.

Our team developed and piloted a novel intervention entitled, Stepped Care to Optimize PrEP Effectiveness in Pregnant and Postpartum women (SCOPE-PP) that addresses barriers to taking daily PrEP by reducing clinic visit frequency and empowering women to adhere to PrEP. Our team will evaluate SCOPE-PP in a pragmatic RCT of pregnant and postpartum women at risk of HIV acquisition. The study will enroll 750 pregnant women in antenatal care and follow them through 12-months' postpartum. Women in the intervention will be offered rapid PrEP collection with enhanced adherence counseling. Women with poor PrEP continuation and/or adherence who want to continue on PrEP will be offered a differentiated care model of PrEP delivery to de-link PrEP from clinical visits. The primary outcome is PrEP continuation and adherence in postpartum women, measured through drug levels of tenofovir diphosphate. The study aims to: 1) Evaluate the efficacy of the SCOPE-PP intervention on PrEP adherence in pregnant and postpartum women in a RCT; 2) Assess the acceptability and feasibility of integrating SCOPE-PP into ante- and postnatal care using a consolidated framework for implementation research (CFIR); and 3) Estimate the incremental cost effectiveness of SCOPE-PP vs. standard of care per HIV infection and disability-adjusted life-year averted. This research is critical to inform maternal PrEP interventions to eliminate HIV acquisition and transmission.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 years
2. Plans to deliver at the study facility
3. Documented HIV-negative according to two finger prick rapid tests (per national protocol for routine antenatal care) and confirmed with a 4th generation antigen HIV test
4. Lives within 20 kilometers of the study facility
5. Without psychiatric or medical contraindications to PrEP use
6. >20 weeks pregnant
7. Able and willing to consent to study participation.

Exclusion Criteria:

Individuals not meeting the above criteria will be excluded.

-

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to PrEP at 6 months after PrEP initiation | 6 months following study enrollment
  Number and proportion of participants who have objective levels of PrEP adherence after 6 months using urine tenofovir test (rapid test of tenofovir, a metabolite of PrEP; yes/no) and blood test (dried blood spots measuring tenofovir diphosphate; categorical measure) comparing the intervention to standard of care arms.
Adherence to PrEP at 15 months after PrEP initiation | 15 months following study enrollment
  Number and proportion of participants who have objective levels of PrEP adherence after 15 months using urine tenofovir test (rapid test of tenofovir, a metabolite of PrEP; yes/no) and blood test (dried blood spots measuring tenofovir diphosphate; categorical measure) comparing the intervention to standard of care arms.

SECONDARY OUTCOMES:
HIV incidence (maternal and infant) | Any time during study follow up (through 15 months after enrollment)
  Number of new HIV infections in women and infants by study arm (diagnosed in study or found in participant medical records)
Adverse events | Any time during study follow up (through 15 months after enrollment)
  Number of participants with adverse events as assessed by CTCAE v4.0, by study arm and treatment exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Gugulethu Midwife Obstetric Unit, Cape Town, South Africa, South Africa

IPD SHARING:
Plan to Share IPD: Yes
The study team will share de-identified data upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year following study start through 1 year following study end
Access Criteria: Email PI with full request: dvoradavey@ucla.edu

REFERENCES:
- [Derived] Joseph Davey DL, Dovel K, Cleary S, Khadka N, Mashele N, Silliman M, Mvududu R, Nyemba DC, Coates TJ, Myer L. Stepped care to optimize pre-exposure prophylaxis (PrEP) effectiveness in pregnant and postpartum women (SCOPE-PP) in South Africa: a randomized control trial. BMC Public Health. 2022 Jul 7;22(1):1306. doi: 10.1186/s12889-022-13652-5. PMID 35799121